CLINICAL TRIAL: NCT04312607
Title: Value of CD26 Positive Stem Cell Marker in Patients With Classical Myeloproliferative Neoplasms
Brief Title: Value of CD26 Positive Leukemic Stem Cell in Myeloproliferative Neoplasm
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Safaa AA Khaled (Other)
Responsible Party: Sponsor-Investigator, Safaa AA Khaled, Value of CD26 positive stem cell marker in patients with classical myeloproliferative neoplasms, Assiut University
Organization: Assiut University (Other)
Other Study IDs: CD26 in MPN
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Myeloproliferative Neoplasm
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Philadelphia chromosome positive: according to PCR detection of BCR-ABL gene CD26 expression on stem cells
  Interventions: Diagnostic Test: BCR-ABL gene PCR
- Philadelphia chromosome negative: according to PCR detection of BCR-ABL gene CD26 expression on stem cells
  Interventions: Diagnostic Test: BCR-ABL gene PCR

INTERVENTIONS:
Diagnostic Test: BCR-ABL gene PCR — peripheral blood sampling for detection of Philadelphia chromosome and flowcytometry for detection of CD26 positive stem cells
  Other Names: flowcytometry for CD26 positive stem cells

SUMMARY:
Evaluate diagnostic and prognostic value of CD26 positive stem cell Stem Cells in classic myeloproliferative neoplasms (MPNs).

To study CD26 expression on different phases of CML (chronic phase, accelerated phase, blastic phase).

To investigate whether CD26 positive stem cell are expressed only in Philadelphia chromosome positive MPN (CML) and/or in Philadelphia chromosome negative MPN (PV, ET, PMF).

DETAILED DESCRIPTION:
Classic Myeloproliferative neoplasms (MPNs) are a heterogeneous group of diseases including Chronic myeloid leukemia (CML), polycythemia vera (PV), essential thrombocythemia (ET), and primary myelofibrosis (PMF) (Levine et al., 2007).

According to WHO 2016 classification which also included chronic neutrophilic leukemia (CNL), chronic eosinophilic leukemia (CEL), and MPN, unclassifiable, Out of the four classic types of MPNs, CML is positive for BCR-ABL1gene , while PV, ET, and PMF are negative for BCR-ABL1 gene (Thapa and Rogers, 2019).

CML is characterized by a balanced genetic translocation, t(9;22)(q34;q11.2), involving a fusion of the Abelson gene (ABL1) from chromosome 9q34 with the breakpoint cluster region (BCR) gene on chromosome 22q11.2. This rearrangement is known as the Philadelphia chromosome, The molecular consequence of this translocation is the generation of a BCR-ABL1 fusion oncogene, which in turn translates into a BCR-ABL oncoprotein (Jabbour and Kantarjian, 2016).

The frontline therapy for patients with CML in chronic phase is tyrosine kinase inhibitors (TKIs) which directed against tyrosine kinase protein of BCR-ABL1 gene. It showed remarkable efficacy and high rates of cytogenetic response in the treatment of chronic phase CML (Yurttaş and Eşkazan, 2020).

However, drug resistance towards tyrosine kinase inhibitors soon emerged and hence limited the complete eradication of CML in patients receiving TKIs. This is primarily due to the mutations within the ABL kinase domain, and to a lesser degree, due to residual disease after treatment (Patel et al., 2018).

Dipeptidyl peptidase IV (DPPIV/CD26) is a transmembrane glycoprotein which has been proposed as an important tumor biomarker in different types of cancer, like melanoma, lung cancer, prostate cancer, gastric and colorectal cancer (Liang et al., 2017) .

CD26 expression in hematological malignancies has been widely studied. It was described as a marker of aggressiveness in T cell malignancies, such as T-acute lymphoblastic leukemias (T-ALL),and associated with poor prognosis and survival ,also found variable expression of CD26 in B cell chronic lymphocytic leukemia (B-CLL) (Enz et al., 2019).

Identification and characterization of leukemic stem cells (LSCs) in CML are one of the recently used investigations. These cells reside within the CD34 positive /CD38 negative and score positive for CD26 which is a marker, expressed in both bone marrow (BM) and peripheral blood (PB) samples, that discriminates CML cells from normal hematopoietic stem cells (HSCs) or from LSCs of other myeloid neoplasms (Raspadori et al., 2017).

the percentage of CD26 LSCs is significantly reduced to low or undetectable levels in CML patients who respond to TKI therapy; however, the percentage of CD26 LSCs remains at high levels in TKI-non responder patients and in patients who have relapsed after TKI therapy, indicating that CD26 could be a useful predictive biomarker for monitoring TKI treatment in CML patients (Raspadori et al., 2019).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed one of classic MPNs (CML, PV, ET, PMF).

Exclusion Criteria:

* Patients below 18 years.
* Pregnancy.
* Any associated Solid or hematopoietic neoplasm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients newly diagnosed one of MPNs for further investigations by PCR for Philadelphia chromosome and flowcytometry for CD26 positve stem cells
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
diagnostic value | within 4 months from study start
  diagnostic value of CD 26 in MPNs

SECONDARY OUTCOMES:
prognostic value | 6 month after start of study
  prognostic value of CD 26 in MPNs

CONTACTS AND LOCATIONS:
Overall Officials: doha M ali, MD, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levine RL, Pardanani A, Tefferi A, Gilliland DG. Role of JAK2 in the pathogenesis and therapy of myeloproliferative disorders. Nat Rev Cancer. 2007 Sep;7(9):673-83. doi: 10.1038/nrc2210. PMID 17721432
- [Background] Thapa B, Fazal S, Parsi M, Rogers HJ. Myeloproliferative Neoplasms. 2023 Aug 8. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK531464/ PMID 30285359
- [Background] Jabbour E, Kantarjian H. Chronic myeloid leukemia: 2016 update on diagnosis, therapy, and monitoring. Am J Hematol. 2016 Feb;91(2):252-65. doi: 10.1002/ajh.24275. PMID 26799612
- [Background] Raspadori D, Pacelli P, Sicuranza A, Abruzzese E, Iurlo A, Cattaneo D, Gozzini A, Galimberti S, Barate C, Pregno P, Nicolosi M, Sora F, Annunziata M, Luciano L, Caocci G, Moretti S, Sgherza N, Fozza C, Russo S, Usala E, Liberati MA, Ciofini S, Trawinska MM, Gozzetti A, Bocchia M. Flow Cytometry Assessment of CD26+ Leukemic Stem Cells in Peripheral Blood: A Simple and Rapid New Diagnostic Tool for Chronic Myeloid Leukemia. Cytometry B Clin Cytom. 2019 Jul;96(4):294-299. doi: 10.1002/cyto.b.21764. Epub 2019 Feb 3. PMID 30714299